CLINICAL TRIAL: NCT03429998
Title: Comparative Pilot Study of the Effectiveness of Evolocumab Versus LDL Apheresis in Patients With Hypercholesterolemia
Brief Title: Evolocumab Versus LDL Apheresis in Patients With Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Marían Goicoechea, MD, PhD, Hospital General Universitario Gregorio Marañon
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVOLAFER01
Record Dates: First submitted 2018-01-28; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Hypercholesterolemia
Keywords: cardiovascular risk; evolocumab; LDL-apheresis
MeSH Terms: conditions — Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: Non-controlled intervention study to evaluate the different therapies in the treatment of hypercholesterolemia, in which each patient will be self-controlled. The variables will be analyzed during different phases
  1. Phase LDL apheresis:
  2. evolocumab phase
  3. Combined phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LDL apheresis (Placebo Comparator): LDL apheresis during at least one year
  Interventions: Procedure: LDL apheresis
- Evolocumab (Active Comparator): 140 mg evolocumab biweekly
  Interventions: Drug: evolocumab
- LDL apheresis and evolocumab (Active Comparator): LDL-apheresis monthly evolocumab 140 mg biweekly
  Interventions: Drug: evolocumab and LDL apheresis

INTERVENTIONS:
Drug: evolocumab — evolocumab 140 mg/biweekly
  Arms: Evolocumab
Drug: evolocumab and LDL apheresis — evolocumab 140 mg/biweekly LDL-apheresis monthly
  Arms: LDL apheresis and evolocumab
Procedure: LDL apheresis — LDL apheresis biweekly
  Arms: LDL apheresis

SUMMARY:
An open-label, prospective phase III study to compare the efficacy and safety of administering evolocumab versus treatment with LDLapheresis in patients with familial hypercholesterolemia and high cardiovascular risk.

DETAILED DESCRIPTION:
STUDY DESIGN An open-label, prospective phase III study to compare the efficacy and safety of administering evolocumab versus treatment with LDLapheresis in patients with familial hypercholesterolemia and high cardiovascular risk.

STUDY POPULATION The chosen population is constituted by patients belonging to the LDL-apheresis program of the General University Hospital Gregorio Marañón with the diagnosis of familial hypercholesterolemia and a history of cardiovascular disease.

Number of patients expected to participate in the study according to the base of patients treated with LDL-apheresis: 10.

STUDY DESIGN:

Non-controlled intervention study to evaluate the different therapies in the treatment of hypercholesterolemia, in which each patient will be self-controlled. The variables will be analyzed during different phases

1. LDL-apheresis phase: Retrospectively during the previous year, pre- and postapheresis variables will be collected from the following lipid parameters: total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, atherogenicity index, Lipoprotein A, apo-A, apo- B; inflammatory parameters: PCR, ferritin, fibrinogen, leukocytes and polymorphonuclear and immunological parameters: immunoglobulins and complement.
2. Evolocumab phase: LDL-apheresis will be suspended for three months and Evolocumab administered: 140 mg / 15 days subcutaneously. The same parameters indicated in the previous section will be measured every two weeks.
3. Combined phase: During the following three months evolocumab will continue to be administered biweekly and the LDL-apheresis procedure will be spaced from biweekly to monthly, the same analytical parameters being measured again every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients with age> 18 years
* hypercholesterolemia with LDL-cholesterol> 100 mg / dl in treatment with the maximum dose tolerated by statins and a history of severe cardiovascular disease
* patients who are included in the LDL-apheresis / biweekly program

Exclusion Criteria:

* contraindications to receive evolocumab according to technical data.
* hospital admission of any cause in the last three months prior to the inclusion of the study
* cardiovascular event in the three months prior to the inclusion of the study
* Inability to sign informed consent
* pregnant women and non-menopausal women who do not use at least one adequate contraceptive method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2018-01-28 (Actual)

PRIMARY OUTCOMES:
decrease in LDL-cholesterol (mg/dl) | 9 months
  decrease in LDL-cholesterol levels in all three phases: LDL-apheresis, evolocumab and combined

SECONDARY OUTCOMES:
Decrease apo-B (mg/dl) levels | 9 months
  decrease in Apolipoprotein B levels in all three phases
Decrease lipoprotein A (mg/dl) levels | 9 months
  decrease in lipoprotein A levels in all three phases
Decrease in triglycerides (mg/dl) levels | 9 months
  Decrease in triglycerides levels in all three phases
any adverse effects | 9 months
  any serious adverse effects
Modification of C reactive protein | 9 months
  Effect of evolocumab and LDL-apheresis on C reactive protein levels (mg/l)
Modification of immunoglobulin G levels (mg/dl) | 9 months
  Effect of of evolocumab and LDL-apheresis on immunoglobulin (mg/dl)
Modification of immunoglobulin A levels (mg/dl) | 9 months
  Effect of evolocumab and LDLapheresis on immunoglobulin A (mg/dl)
Modification of complement levels (mg/dl) | 9 months
  Effect of evolocumab and LDL apheresis on serum complement (mg/dl)
Modification of serum fibrinogen (mg/dl) | 9 months
  Effect of evolocumab and LDL-apheresis on serum fibrinogen (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Marian Goicoechea, MD, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañon
Locations (1):
- Hospital General Universitario Gregorio Marañon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No